CLINICAL TRIAL: NCT02323503
Title: BIOtronik Study to Assess the CONTINUation of Existing Risk of Ventricular Arrhythmias After CRT-D Replacement for Patients With Primary Prevention Indication
Brief Title: Assessment of Ventricular Arrhythmia Risk After CRT-D Replacement for Patients With Primary Prevention Indication
Acronym: BioCONTINUE
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: CR018
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2019-06

CONDITIONS: Cardiac Resynchronization; Biventricular Pacemakers, Artificial; Cardioverter-Defibrillators, Implantable; Device Replacement
Keywords: CRT-D; replacement; primary prevention; ventricular tachyarrhythmias
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CRT-D device replacement

SUMMARY:
Cardiac resynchronization therapy (CRT) has been shown to reduce heart failure (HF), hospitalizations and death in patients with left ventricular ejection fraction (LVEF) <35% and wide QRS. CRT provides electromechanical resynchronization and improves LV systolic function. The induced LV reverse remodeling or near normalization in LVEF to ≥45% is associated with a significant reduction in the risk of subsequent life-threatening ventricular tachyarrhythmias (VTA). And at the time of replacement, the need for defibrillator back-up after an event-free first CRT-D service-life for patients with improved LVEF is a controversy question.

80% of Implantable Cardioverter Defibrillator (ICD) patients implanted for primary prevention do not experience VTA during the life-time of their first device.

So, regarding patients implanted with a CRT-D for primary prevention at the time of first implantation, the question is will they experience VTA after their device replacement by another CRT-D.

DETAILED DESCRIPTION:
The objective of this study is to describe, in a population of patients who had a primary prevention ICD indication at first implantation of a CRT-D, the relevance defibrillator back-up after the replacement of the first CRT-D. For that, the rate of patients with at least one sustained VTA detected by the CRT-D or a conventional surface ECG will be assessed after the device replacement.

Furthermore, the association between the baseline characteristics of the CRT-D population after replacement and the risk of subsequent VTA will be explored after a minimum of two years FU.

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary prevention indication for defibrillation at the time of the first CRT-D implantation
* Patient implanted as first replacement by a CRT-D device (CRT-D by CRT-D)
* Lifetime of the previous CRT-D > 3 years
* Patient willing and able to comply with the protocol and who has provided written informed consent
* Patient whose medical situation is stable.

Exclusion Criteria:

* Patient with an ICD lead under advisory (e.g. Fidelis lead)
* Right or left ventricular leads exchange during CRT-D replacement
* Non functional atrial (except for patient with chronic AF) or right/left ventricular leads
* Life expectancy < 1 year
* Age < 18 years
* Pregnant woman or woman who plan to become pregnant during the trial
* Participation in another interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients initially implanted with a CRT-D (cardiac resynchronization therapy with defibrillator) device for primary prevention indication for defibrillation, requiring a device replacement by another CRT-D because of battery depletion
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Assess the rate of patients with at least one sustained VTA after replacement | up to two years

SECONDARY OUTCOMES:
Rate of patients with at least one VTA for 4 specific subgroups | After the device replacement and after a minimum of two years follow-up (FU)
  Grp R[1-4]: LVEF ≥40% / <40% at the time of replacement and with / without previous VTA during the lifetime of their first CRT-D device

OTHER OUTCOMES:
Rate of patients with ventricular tachycardia or ventricular fibrillation events, with appropriate therapies | After the device replacement and after a minimum of two years FU
Rate of patients with inappropriate therapies/diagnosis | After the device replacement and after a minimum of two years FU
Baseline factor predictors of ventricular events | After the device replacement and after a minimum of two years FU
Serious adverse events related to ventricular events / inappropriate therapies | After the device replacement and after a minimum of two years FU

CONTACTS AND LOCATIONS:
Overall Officials: Daniel DG Gras, MD, Principal Investigator — Nouvelles Cliniques Nantaises, France
Locations (37):
- OLV Aalst, Aalst, Belgium
- France (22):
  - CH d'Annecy, Annecy
  - Hôpital de la Cavale Blanche, Brest
  - CHU Caen, Caen
  - CHU Montpied, Clermont-Ferrand
  - CH Du Bocage, Dijon
  - CHRU de Lille, Lille
  - CHU de Limoges, Limoges
  - CH Saint Philibert, Lomme
  - Cliniques du Tonkin, de la Sauvegarde et Protestante, Lyon
  - Clinique Clairval, Marseille
  - Hôpital de la Timone, Marseille
  - Hôpital Mercy, Metz
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - Nouvelles Cliniques Nantaises, Nantes
  - CH de la Pitié Salpétrière, Paris
  - CHU Pessac, Pessac
  - CHU de Rennes, Rennes
  - CHU Hôpital CHarles Nicolle, Rouen
  - CH de Saint-Etienne, Saint-Etienne
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
- Germany (4):
  - Schuechtermann-Klinik, Bad Rothenfelde
  - Stadtisches Klinikum Brandenburg, Brandenburg
  - DRK-Krankenhaus Moelln Ratzeburg, Ratzeburg
  - Cardiological Praxis, Rostock
- Semmelweis University, Budapest, Hungary
- Barzilai Medical Center, Ashkelon, Israel
- Italy (3):
  - Ospedale Versilia, Lido di Camaiore
  - Clinica Mediterranea, Napoli
  - Ospedale Santa Chiara, Pisa
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - Hospital de Santa Marta, Lisbon
- Spain (3):
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gras D, Clementy N, Ploux S, Guyomar Y, Legallois D, Segreti L, Blangy H, Laurent G, Bizeau O, Fauquembergue S, Lazarus A; BioCONTINUE study Investigators. CRT-D replacement strategy: results of the BioCONTINUE study. J Interv Card Electrophysiol. 2023 Aug;66(5):1201-1209. doi: 10.1007/s10840-022-01440-5. Epub 2022 Dec 2. PMID 36459310